CLINICAL TRIAL: NCT01386476
Title: The Serotonin-1A Receptor Radioligand (18F)FCWAY as a Potential Substrate for Efflux Transport at the Blood-Brain Barrier
Brief Title: (18F)FCWAY and the Blood-Brain Barrier
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110195; 11-M-0195
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-09-01

CONDITIONS: Drug Resistance
Keywords: 5-HT1A Receptors; Blood Brain Barrier; Drug Resistance; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- The blood-brain barrier helps protect the brain from infections and toxins in the blood stream. But it can also prevent certain drugs from reaching the brain to treat diseases or other problems. Researchers are interested in chemicals that will help show how the barrier works. One possible chemical, (18F)FCWAY, may be useful for studying the barrier. More tests are needed to determine how effective it is.

Objectives:

- To test whether (18F)FCWAY can be used to help study the blood-brain barrier.

Eligibility:

- Healthy volunteers between 18 and 50 years of age.

Design:

* This study requires a screening visit and two scanning visits.
* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests.
* At the first scanning visit, participants will have a magnetic resonance imaging scan to provide baseline images of the brain.
* Before the second visit, some participants will stay overnight in the hospital. They will receive the drug tariquidar, which may help the (18F)FCWAY show the blood-brain barrier more clearly.
* At the second scanning visit, all participants will have a positron emission tomography scan with (18F)FCWAY to see how well the drug shows the blood-brain barrier on the scan.

DETAILED DESCRIPTION:
Objective:

We use the radioligand [(11)C]dLop (N-desmethyl-loperamide) in positron emission tomography (PET) studies to measure function of P-gp, an efflux transporter at the blood-brain barrier. Because [(11)C]dLop is an avid substrate for P-gp, we see almost no radioactivity in brain at baseline in healthy volunteers. However, we do see increased radioactivity in brain in some patients with dementia, or when we co-administer a medication which blocks the function of P-gp. While [(11)C]dLop is useful for detecting increased radioactivity in brain, a disadvantage of [(11)C]dLop is that it is not useful for detecting decreased radioactivity in brain. The reason for this is that we have a floor effect, where we are unable to detect less radioactivity than zero. Preclinical studies indicate that increases in P-gp activity (which would manifest as decreased radioactivity in brain) correlate with drug-resistant epilepsy and HIV. To better understand diseases associated with not only increased but also decreased P-gp activity, we wish to identify a radioligand which is a moderate substrate of P-gp. We suspect that [(18)F]FCWAY is a moderate substrate for P-gp, because some radioligand gets into brain at baseline, but more gets into brain after administering a drug (disulfiram) which inhibits P-gp. The objective of this study is to determine whether the serotonin 1A antagonist [(18)F]FCWAY is a substrate of P-gp by determining whether the P-gp inhibitor, tariquidar, increases uptake of the radioligand into brain.

Study Population:

We will study up to 45 healthy adults, ages 18-50. Participants must be free of medications, with the exception of birth control pills, as medications may confound our data. or iii patients who received a single PET scan as stated under i), will be invited back to have the option of receiving the second PET scan with tariquidar. A maximum of 15 ubjects will receive both scans.

Design:

Healthy adults will undergo either 1) a single PET scan of the brain with [(18)F]FCWAY (at baseline, or during infusion of intravenous tariquidar or 2) two PET scans (both a baseline and a tariquidar scan).

Outcome Measures:

If [(18)F]FCWAY is a substrate of P-gp, pre-treatment with tariquidar will increase its brain uptake of [(18)F]FCWAY and delay the time of peak uptake.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be 18 to 50 years old.

Subjects must be currently healthy, based on history, physical exam, and laboratory testing.

With the exception of birth control pills, subjects must agree not to take any medication, prescription or over-the-counter, one week before and one week after receiving tariquidar.

Subjects must be able and willing to give written informed consent.

EXCLUSION CRITERIA:

Subjects routinely taking prescription medications, except birth control pills. That is, subjects should not discontinue mediations merely to participate in this study.

Subjects taking recreational or over-the-counter drugs.

Subjects will be excluded if they have any current Axis I diagnosis, including a current diagnosis of alcohol or substance abuse.

History of psychotic symptoms or suicide attempt.

Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes or a history of seizures, because seizures may increase the function of P-gp.

Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.

Pregnancy or breast feeding.

Positive urine drug screen.

Unlikely to tolerate small, enclosed spaces, as in the MRI.

Metallic foreign bodies that would be affected by the MRI magnet or fear of enclosed spaces likely to make the subject unable to complete an MRI scan.

Positive HIV status.

Inability to lie flat on camera bed for about 2 (Omega) hours.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06-15; Study Completion 2016-09-01

PRIMARY OUTCOMES:
Tariquidar will increase uptake of 18F-FCWAY in brain

SECONDARY OUTCOMES:
Tariquidar will delay brain peak of 18F-FCWAY

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kannan P, John C, Zoghbi SS, Halldin C, Gottesman MM, Innis RB, Hall MD. Imaging the function of P-glycoprotein with radiotracers: pharmacokinetics and in vivo applications. Clin Pharmacol Ther. 2009 Oct;86(4):368-77. doi: 10.1038/clpt.2009.138. Epub 2009 Jul 22. PMID 19625998
- [Background] Zhang XY, Yasuno F, Zoghbi SS, Liow JS, Hong J, McCarron JA, Pike VW, Innis RB. Quantification of serotonin 5-HT1A receptors in humans with [11C](R)-(-)-RWAY: radiometabolite(s) likely confound brain measurements. Synapse. 2007 Jul;61(7):469-77. doi: 10.1002/syn.20392. PMID 17415792
- [Background] Liow JS, Lu S, McCarron JA, Hong J, Musachio JL, Pike VW, Innis RB, Zoghbi SS. Effect of a P-glycoprotein inhibitor, Cyclosporin A, on the disposition in rodent brain and blood of the 5-HT1A receptor radioligand, [11C](R)-(-)-RWAY. Synapse. 2007 Feb;61(2):96-105. doi: 10.1002/syn.20348. PMID 17117422